CLINICAL TRIAL: NCT02745834
Title: The Influence of Dual Task and Gait Speed on Gait Variability in Patients With Chronic Ankle Instability - a Case-control Study
Brief Title: The Influence of Dual Task and Gait Speed on Gait Variability in Patients With Chronic Ankle Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Collaborators: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IDF-1482-2014
Record Dates: First submitted 2016-03-15; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Instability of Joint
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Ankle Instability (Experimental): Soldiers who suffer from chronic ankle instability who had a first major ankle sprain one year or more ago, and did not sustained any major ankle sprain in the last two months, will go through Gait analysis intervention.
  Interventions: Other: Gait analysis
- Healthy controls (Experimental): Healthy soldiers who are not suffering from chronic ankle instability, will go through Gait analysis intervention.
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — Gait will be analysed while participants will walk on a treadmill at different self selected speeds, using the OPTOGait system. Spatiotemporal measures are collected without the use of any markers.

SUMMARY:
Case-control study to evaluate gait parameters during different conditions between patients who suffer from chronic ankle instability and healthy individuals.

DETAILED DESCRIPTION:
This case-control study will compare the different gait parameters such as stride time and stride length variability in different gait conditions (e.g., normal speed, normal speed with dual task, fast speed and fast speed with dual task) between healthy individuals and patients who suffer from chronic ankle instability.

the measurements will be collected using the OPTOGait system installed on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

* history of at least one significant ankle sprain which occurred at least 12 months prior to enrolment in the study and was diagnosed by a physician or a physical therapist using clinical examination classifications described by Malliaropoulos et al
* history of at least two episodes of 'giving way', and feelings of ankle joint instability in the previously injured ankle joint of 1 year post-initial sprain
* the most recent injury occurred more than 6 weeks prior to the study enrolment
* the ability to apply full weight bearing on the injured lower extremity with no more than mild discomfort

Exclusion Criteria:

* evidence of a concomitant injury (such as a bony injury or significant muscular/tendon injury)
* previous ankle surgery
* other pathological conditions or surgical procedures in lower extremity
* neurological/vestibular or any other balance disorder.

The control group included healthy participants with no current or previous conditions that could affect proprioception.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Stride time variability | Day 1
  Coefficient of variance of the stride time, measured in % by the OPTOGait system
Stride length variability | Day 1
  Coefficient of variance of the stride length, measured in % by the OPTOGait system

SECONDARY OUTCOMES:
Dual task general score | Day 1
  Participants will be asked to count backward, reducing 7 at a time, starting at different 3 digits number. The outcome measure is a calculation of the number of total answers multiple by (number of correct answers - number of wrong answers).

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Springer, PhD, Principal Investigator — Researcher
Locations (1):
- IDF Medical Corp, Zrifin, Israel

IPD SHARING:
Plan to Share IPD: No
Data will be published after statistical analysis only.

REFERENCES:
- [Derived] Springer S, Gottlieb U. Effects of dual-task and walking speed on gait variability in people with chronic ankle instability: a cross-sectional study. BMC Musculoskelet Disord. 2017 Jul 21;18(1):316. doi: 10.1186/s12891-017-1675-1. PMID 28732483